CLINICAL TRIAL: NCT07286734
Title: Ultrasound Assesment Of Radial Nerve In Humeral Shaft Fracture Patients With Radial Palsy
Status: Recruiting | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Mahmut Gumus, Professor, Istanbul Medeniyet University
Other Study IDs: IstanbulMU_032025
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Humerus Shaft Fracture; Radial Nerve Palsy
MeSH Terms: conditions — Radial Neuropathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radial Nerve Palsy Group: Patients with humeral shaft facture and Radial Nerve Palsy
  Interventions: Device: High-Resolution Ultrasound Evaluation of the Radial Nerve
- No radial Nerve Palsy: Patients with humeral shaft fracture but no radial nerve palsy
  Interventions: Device: High-Resolution Ultrasound Evaluation of the Radial Nerve

INTERVENTIONS:
Device: High-Resolution Ultrasound Evaluation of the Radial Nerve — High-resolution diagnostic ultrasound of the radial nerve is performed using a linear transducer (6-15 MHz) within 48 hours of admission in patients with humeral shaft fractures. The ultrasound systematically assesses the radial nerve's continuity, morphology, and relation to the fracture site. Based on established classification criteria (e.g., stretch neuropraxia, incarceration, partial/complete transection), the ultrasound findings guide intraoperative planning. All imaging is performed by board-certified musculoskeletal radiologists following a standardized protocol.

SUMMARY:
This study investigates how well ultrasound imaging can identify damage to the radial nerve in patients with a broken upper arm bone (humeral shaft fracture). Some of these patients also have weakness or paralysis in their hand and wrist due to injury to the radial nerve. The study compares patients with and without radial nerve problems to see if early ultrasound scans can accurately detect nerve damage before surgery.

All patients will receive standard care, including surgery to fix the fracture. Those with nerve problems will also have the nerve explored during surgery. The results of the ultrasound will be compared to what is found during the operation. Patients will be followed closely over 12 months to monitor nerve recovery, healing of the bone, and any complications.

The goal is to improve the early diagnosis and management of nerve injuries in arm fractures, using a safe, non-invasive ultrasound scan that could help guide treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Diagnosed with traumatic humeral shaft fracture.
* Admitted and followed according to the local clinical protocol with a confirmed diagnosis.
* Underwent required investigations, including high-resolution ultrasonography and/or electromyography (EMG).
* Provided written informed consent to participate in the study.

Exclusion Criteria:

* Pathological fractures due to malignancy or metabolic disorder.
* History of previous humeral fracture or pre-traumatic radial nerve deficit.
* Clinically detected vascular injury or major soft tissue loss accompanying the fracture.
* Incomplete diagnostic workup (absence of ultrasound or EMG examination).
* Declined participation or were lost to follow-up.
* Persons under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting with acute traumatic humeral shaft fractures at a tertiary care orthopedic center. Patients are assigned to cohorts based on the presence or absence of clinical radial nerve palsy. All participants undergo standard diagnostic and therapeutic procedures, with targeted ultrasound used for nerve assessment in the radial palsy group.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Preoperative Ultrasound Accuracy in Detecting Radial Nerve Continuity | Baseline (within 48 hours of admission); confirmation at surgery
  This outcome assesses how accurately high-resolution ultrasonography identifies whether the radial nerve is intact in patients with humeral shaft fractures and radial nerve palsy. The ultrasound findings will be compared to surgical exploration results (reference standard). Diagnostic accuracy metrics include sensitivity, specificity, positive predictive value, and negative predictive value.

SECONDARY OUTCOMES:
Correlation Between Ultrasound Classification and Intraoperative Radial Nerve Findings | Baseline (ultrasound), Intraoperative, and Postoperative (3, 6, and 12 months)
  Ultrasound-based classification of radial nerve injury (e.g., stretch, incarceration, partial/complete transection) will be compared with intraoperative findings to assess diagnostic agreement. Additional analyses will evaluate the relationship between USG classification and postoperative functional outcomes
Functional Recovery of Radial Nerve Motor and Sensory Function | 1, 3, 6, and 12 months postoperatively
  Recovery of motor function (wrist/finger/thumb extension) will be evaluated using the Medical Research Council (MRC) scale (0-5). Sensory recovery will be assessed via light touch and pinprick sensation in the radial nerve territory. Outcomes include proportion of patients with full, partial, or no recovery, and time to initial and full improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No